CLINICAL TRIAL: NCT01265602
Title: Double-blind, Randomized, Vehicle- and Comparator-controlled, Multi-center Trial to Evaluate the Efficacy and Safety of LAS41007 in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H 569 000 - 1004
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; AK; NMSC
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- LAS41007 (Experimental): All patients will be instructed to apply the IMP twice daily, once in the morning and once in the evening. Per application, not more than 1.5 g of the IMP should be applied, which is sufficient to cover a total area of 75 cm2 (corresponding to 3 single TAs, each with a size of 25 cm²) in maximum. The IMPs will be applied for 90 days in maximum.
  Interventions: Drug: LAS41007
- LASW1510 (Active Comparator): All patients will be instructed to apply the IMP twice daily, once in the morning and once in the evening. Per application, not more than 1.5 g of the IMP should be applied, which is sufficient to cover a total area of 75 cm2 (corresponding to 3 single TAs, each with a size of 25 cm²) in maximum. The IMPs will be applied for 90 days in maximum.
  Interventions: Drug: LASW1510
- vehicle (Placebo Comparator): All patients will be instructed to apply the IMP twice daily, once in the morning and once in the evening. Per application, not more than 1.5 g of the IMP should be applied, which is sufficient to cover a total area of 75 cm2 (corresponding to 3 single TAs, each with a size of 25 cm²) in maximum. The IMPs will be applied for 90 days in maximum.
  Interventions: Drug: vehicle of LAS41007

INTERVENTIONS:
Drug: LAS41007 — Topical gel, to be applied twice daily (mornings and evenings), for up to 90 days. Generally 0.5 g gel (pea-sized amount of gel) per application will be sufficient to cover an overall area of 25 cm².
  Arms: LAS41007
Drug: LASW1510 — Topical gel, to be applied twice daily (mornings and evenings), for up to 90 days. Generally 0.5 g gel (pea-sized amount of gel) per application will be sufficient to cover an overall area of 25 cm².
  Arms: LASW1510
Drug: vehicle of LAS41007 — Topical gel, to be applied twice daily (mornings and evenings), for up to 90 days. Generally 0.5 g gel (pea-sized amount of gel) per application will be sufficient to cover an overall area of 25 cm².
  Arms: vehicle

SUMMARY:
The aim of this study is to determine the efficacy, safety and tolerability of LAS41007 compared to a marketed reference product as well as to vehicle (topical application, twice daily, indication mild to moderate AK).

ELIGIBILITY:
Inclusion Criteria:

* Have at least 6 but not more than 16 clinically confirmed AK target lesions of mild to moderate (grade I to II, according to Olsen et al., 1991) intensity in the whole treatment area (TA) (and additionally one representative AK lesion for histological diagnosis of AK), which must be located in the face including the forehead (excluding eyelids, lips and mucosa) and/or bald scalp,
* The AK target lesions must be discrete and quantifiable; the distance from one lesion to its neighbor lesion must be greater than 1.0 cm,
* The diameter of each AK target lesion should be not less than 0.5 cm and not greater than 1.5 cm,
* The target lesions must be located in up to 3 TAs with a size of 25 cm2 per TA (i.e. total area of TA is up to 75 cm2),
* Diagnosis of AK histologically confirmed

Exclusion Criteria:

* Have known hypersensitivity, intolerance or allergies against ingredients of the IMPs and other non-steroidal anti-inflammatory agents,
* Have a history of bronchospasm, asthma, urticaria, or rhinitis after the intake of non-steroidal anti-inflammatory drugs (NSAIDs),
* Have a history of gastrointestinal bleeding or perforation associated with prior therapy with NSAIDs,
* Have evidence of clinically significant or unstable medical conditions,
* Have currently and within the past 3 months other malignant tumors of the skin in the TAs,
* Suffer from paresthesia in the TAs,
* Show cornu cutaneum of the skin and/or hypertrophic AK lesions in the TAs,
* Are known to be pregnant or lactating (currently or within the past 3 months),
* Any clinically relevant abnormal finding during Screening and/or Baseline,
* Specific topical treatments in the target area within defined time periods.
* Specific physical treatments in the TAs within defined time periods.
* Specific systemic treatments within defined time periods.
* Patients suffering from AK in locations other than the target areas, receiving any topical AK-therapy throughout the interventional phase of the study until termination of V6,
* Patients who need a permanent therapy with any other NSAID. The use of NSAIDs as "prn" (pro re nata), i.e. to be taken as needed (≤ 3 days at a stretch) and the use of ASA as anticoagulative therapy will be allowed,
* Patients taking methotrexate or sulfonylurea during the interventional phase of the study,
* Anticoagulative therapy, e.g. with cumarines or heparines throughout the interventional phase of the study. Treatment with ASA at a dose not exceeding 100 mg/d and clopidogrel at a dose not exceeding 75 mg/d will be allowed,
* Patients having any significant physical abnormalities in the potential TAs that may cause difficulty with examination or final evaluation,
* Have any dermatological disease in the TAs or surrounding area that may be exacerbated by treatment with topical diclofenac or cause difficulty with examination,
* Physical or mental inability and/or unwillingness to apply the study preparations correctly and to follow the study restrictions and visits,
* Any suspicion of current drug and/or alcohol abuse as assessed by the investigator,
* Anticipated non-availability for study visits / procedures,
* Exposure to an investigational product within the last 3 months,
* Any previous randomization into this trial,
* Patient is institutionalized because of legal or regulatory order,
* Employee of the study site or of the Sponsor's company or the CRO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
superiority of LAS41007 compared to vehicle | Day 1
  superiority of LAS41007 compared to comparator each assessed by histology to evaluate the histological clearance of one pre-selected target lesion
superiority of LAS41007 compared to vehicle | Day 150
  superiority of LAS41007 compared to comparator each assessed by histology to evaluate the histological clearance of one pre-selected target lesion

SECONDARY OUTCOMES:
superiority of LAS41007 compared to vehicle | Day 1
  improved clinical efficacy of LAS41007 compared to comparator with respect to clinical efficacy
superiority of LAS41007 compared to vehicle | Day 21
  improved clinical efficacy of LAS41007 compared to comparator with respect to clinical efficacy
superiority of LAS41007 compared to vehicle | Day 56
  improved clinical efficacy of LAS41007 compared to comparator with respect to clinical efficacy
superiority of LAS41007 compared to vehicle | Day 90
  improved clinical efficacy of LAS41007 compared to comparator with respect to clinical efficacy
superiority of LAS41007 compared to vehicle | Day 150
  improved clinical efficacy of LAS41007 compared to comparator with respect to clinical efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Estrella Estrella Garcia, PhD, Study Director — Almirall, S.A.
Locations (1):
- Almirall Investigational Site, Vechta, Germany